CLINICAL TRIAL: NCT04991012
Title: Evaluation of the Effectiveness of Photodynamic Therapy in the Treatment of Lesions of the Lichen Planus Type in the Oral Mucosa and Its Diagnostics With the Use of Autofluorescence, in Various Wavelength Ranges, in Combination With the Use of Texture Analysis and Fractal Dimension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kb845/2020
Record Dates: First submitted 2021-06-17; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-06

CONDITIONS: Oral Lichen Planus
Keywords: photodynamic therapy
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Photochemotherapy; Triamcinolone

STUDY DESIGN:
Intervention Model Description: full contralateral split-mouth
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photodynamic therapy side (Experimental): On one side, the OLP lesion eligible for treatment was subjected to photodynamic therapy in four sessions every 2 days.Using as photosensitizer Methylen blue for 10min the lesion was irradiated with a 650 nm semiconductor laser at a dose of 120 J / cm2
  Interventions: Device: PDT Therapy
- Triamcinolone (Substance) therapy side (Active Comparator): on the other side The OLP on the other side was treated by daily sticking a cut-to-size carrier with 0.05% triamcinolone acetonide for 8 days
  Interventions: Drug: Triamcinolone (Substance) therapy side

INTERVENTIONS:
Device: PDT Therapy — the olp was photosensitized with methylen blue and was irradiated with a semiconductor laser with a wavelength of 650 nm, using a dose of 120 J / cm2 and power density
  Other Names: Photodynamic Therapy
  Arms: photodynamic therapy side
Drug: Triamcinolone (Substance) therapy side — th The OLP on the other side was treated by daily sticking a cut-to-size carrier with 0.05% triamcinolone acetonide for 8 days
  Other Names: Steroid therapy
  Arms: Triamcinolone (Substance) therapy side

SUMMARY:
Lesions of the lichen planus type within the oral mucosa are now considered a potentially cancerous condition. One of the minimally invasive methods of treating these lesions is photodynamic therapy, and the gold standard in therapy is topical steroid administration

DETAILED DESCRIPTION:
Lichen planus shows an irregular shape, which is quite difficult to measure objectively, which is important in assessing the effectiveness of treatment.

Patients will be treated in protocol split mouth with the treatment of lesions on one cheek with a steroid (on an adhesive plaster) and on the other - photodynamic therapy with a foot sensitizer in the form of a methylene blue also on an adhesive plaster The treatment evaluation procedure will consist of taking a series of intraoral photographs. These photos will be taken at each visit. This procedure will involve taking pictures traditionally in "white" light and in the spectrum of 405 nm, 460 nm and 405 + 460 nm (using the unique feature of the prototype laser - emission of two wavelengths simultaneously) in order to induce autofluorescence of the mucosa and treated lesions to better visualize them

A prospective, randomized, single-blind 12-week clinical trial of full contralateral split-mouth in patients with bilateral erythematous or erosive lichen planus in the mouth.On one side, the OLP lesion eligible for treatment was subjected to photodynamic therapy using methylene blue in four sessions every 2 days.

olp on the other side was treated with the administration of the steroid triamcinolone for 8 days

The clinical evaluation of the evolution of OLP eruptions was performed within 12 weeks of qualifying for treatment: at baseline, at the end of both treatments (day 8) and after the next 11 weeks

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of OLP
* non smoker
* no diabetes melitus
* no hepatitis

Exclusion Criteria:

* diabetes melitus
* hepatitis
* occurrence dysplasia in the histopathological specimen;
* use of lichenoid reaction inducing medication and presence of amalgam fillings nearby the lesions;
* interventions for OLP in the previous 12 weeks;
* pregnant or breastfeeding women;
* proved or suspected hypersensitivity to any of the chemicals used in the treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
length of oral lichen planus | 12 weeks
  The measurement was made with a periodontal probe PCP UNC 15 in millimeters
  we measured the length of the lesions
height of oral lichen planus | 12 weeks
  The measurement was made with a periodontal probe PCP UNC 15 in millimeters
  we measured the height

SECONDARY OUTCOMES:
computer analysis of autofluorescence of lesions | 12 weeks
  Based on photos taken in various light spectrum and fractal analysis of changes
  In this study, we used two wavelengths: 405, 450 and 405+450 nm together for the autofluorescence of lesions
  All fractal analysis was performed in ImageJ version 1.53e (Image Processing and Analysis in Java)
  Applied the intensity difference fractal dimension counting method.
  We measured the size of oral lichen planus on photos taken with different light wave using computer program as mentioned above

CONTACTS AND LOCATIONS:
Overall Officials: kamil jurczyszyn, prof, Study Director — Wroclaw Medical University; tomasz konopka, prof, Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No